CLINICAL TRIAL: NCT02750228
Title: Patent Ductus Arteriosus Post NICU Discharge in Premature Infants: A Prospective Registry
Brief Title: PDA Post NICU Discharge
Acronym: PDA
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-002-15
Record Dates: First submitted 2016-03-23; First posted 2016-04-25 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to track post-discharge outcomes on prematurely born infants who are discharged from the NICU with a patent ductus arteriosus (PDA). Investigators plan to report on the spontaneous closure rate as well as the incidence of pulmonary and/or cardiac events in these infants. The goal is to identify risk factors associated with adverse outcomes in prematurely born infants who are sent home with a PDA.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of informed consent and authorization for participation.
* Estimated gestational age of 32 weeks or less.
* Active diagnosis of a PDA at discharge.
* At least one echocardiogram obtained during hospital stay documenting/ confirming PDA diagnosis.
* Parental agreement to provide follow-up information on their child.
* Cardiologist and/or Pediatrician willing to provide follow-up information on enrolled infants.

Exclusion Criteria:

* No known major congenital anomalies (inborn error of metabolism, cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia or other major gastrointestinal anomalies, major neurological injury or anomaly, multiple congenital anomalies).
* Chromosomal / genetic disorders - Inherited metabolic disorders (Aa, fat or carbohydrate), Trisomies, Turner's syndrome,Vater's syndrome, CHARGE, DiGeorge or other 22q11 deletions, Major chromosomal duplications, deletions detectable on high resolution karyotype (not microarray).
* Parent(s) unwilling to participate in follow-up.

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a prospective multicenter descriptive study to collect data on neonatal outcomes and treatment modalities of neonates diagnosed with a patent ductus arteriosus by echocardiogram and have an active diagnosis of a PDA at discharge from the hospital.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2016-05; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects that have a report of a spontaneous closure of PDA, medication intervention for closure of PDA or surgical intervention for closure of PDA | 18 months

SECONDARY OUTCOMES:
Number of subjects with or without a closure of PDA that have heart failure, pulmonary arterial hypertension, a need for respiratory support and death | 18 months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Winnie Palmer Hospital for Women & Babies, Orlando, Florida
  - MEDNAX Center for Research, Education and Quality, Sunrise, Florida
  - Northside Hospital, Atlanta, Georgia
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Greenvillle Memorial Hospital, Greenville, South Carolina
  - Seton Medical Center, Austin, Texas
  - Dell Children's Medical Center, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital, San Antonio, Texas
  - Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Derived] Tolia VN, Powers GC, Kelleher AS, Walker MW, Herrman KK, Ahmad KA, Buchh B, Egalka MC, Hinkes M, Ma M, Richards M, Rudine AC, Sato RY, Shaffer KM, Clark RH. Low Rate of Spontaneous Closure in Premature Infants Discharged with a Patent Ductus Arteriosus: A Multicenter Prospective Study. J Pediatr. 2022 Jan;240:31-36.e2. doi: 10.1016/j.jpeds.2021.07.035. Epub 2021 Jul 20. PMID 34293369